CLINICAL TRIAL: NCT07172672
Title: Impact of Meal Insulin Dose Timing on Meal Fat Storage in Patients With Type 1 Diabetes: a Randomized Control Trial - the TiMeD-T1D Project
Brief Title: The TiMeD-T1D Project
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: TiMed-T1D
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Postprandial Lipid Metabolism; Type 1 Diabetes (T1D)
Keywords: FTHA PET; Insulin; Postprandial metabolism; Human; Meal fat storage in skeletal muscle, liver, brain, and subcutaneous fat adipose tissue
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meal insulin bolus 20 min before consumption of a liquid mixed meal (Experimental)
  Interventions: Dietary Supplement: 400 mL Fresubin Energy Drink and 100 mL heavy cream with the addition of the 18F-FTHA radiotracer
- Meal insulin bolus 20 min after consumption of a liquid mixed meal (Experimental)
  Interventions: Dietary Supplement: 400 mL Fresubin Energy Drink and 100 mL heavy cream with the addition of the 18F-FTHA radiotracer
- Skipping the insulin bolus (Experimental)
  Interventions: Dietary Supplement: 400 mL Fresubin Energy Drink and 100 mL heavy cream with the addition of the 18F-FTHA radiotracer

INTERVENTIONS:
Dietary Supplement: 400 mL Fresubin Energy Drink and 100 mL heavy cream with the addition of the 18F-FTHA radiotracer — 400 mL Fresubin Energy Drink and 100 mL heavy cream with the addition of the 18F-FTHA radiotracer

SUMMARY:
The aim of the proposed study is to investigate the metabolic consequences of varying the timing of meal insulin boluses and skipping boluses altogether in individuals with type 1 diabetes.

The investigator hypothesize that delaying or skipping meal insulin boluses leads to greater ectopic fat storage due to a delayed stimulation of lipoprotein activity and delayed suppression of lipolysis and VLDL-TG secretion.

DETAILED DESCRIPTION:
The study will be carried out as a randomized cross-over clinical investigational trial. The investigators will include 10 individuals with type 1 diabetes. The subjects will be invited for four visits in total: one screening visit and three test days separated by a one-week washout period. At the test days, subjects will consume a liquid mixed meal and: 1) take a meal bolus of insulin 20 min before consuming a liquid mixed meal or 2) take a meal bolus of insulin 20 min after the meal or 3) skip the meal bolus of insulin.

The investigators will apply the 18F-FTHA meal fat tracer method to the liquid mixed meal to determine whole-body organ-specific meal fat storage.

The volunteers will arrive fasted (8 hours) at the Department of Nuclear Medicine & PET-Centre at 9.00 a.m. Upon arrival, participants will be placed in a bed and have an arterial catheter placed for arterial blood sampling collected at baseline and during the entire trial day. Approximately one hour after arriving, participants will consume a liquid mixed meal consisting of 400 mL Fresubin Energy Drink and 100 mL heavy cream with the addition of the 18F-FTHA radiotracer. 5 hours after consumption of the liquid mixed meal one static whole-body PET-scan will be performed with a duration of 1 hours. After the PET-scan participants will be provided with a meal. Subsequently, the investigator will make sure the participants is metabolic corrected and then the trial day is ended, and they can go home.

The three test days will be conducted in the same way, except for the timing of insulin bolus administration relative to the meal, which will vary as follows:

1. Meal insulin bolus 20 min before consumption of a liquid mixed meal (as recommended)
2. Meal insulin bolus 20 min after consumption of a liquid mixed meal
3. Skipping the insulin bolus Insulin will be administered subcutaneously, with the dose determined based on the composition of the liquid mixed meal.

To correct for attenuation, the investigators will perform one ultra-low dose, non-contrast enhanced CT scan on each study day.

Results will be presented as means ± SD when possible. Primary and secondary outcomes will be analyzed using a two-way mixed model of linear regression with repeated measurements together with standard statistical methodology to compare results between study days. P-values < 0.05 will be considered statistically significant. Statistical analyses will be carried out using R and visualization with GraphPad Prism.

The investigators base the sample size on our primary endpoint visceral meal fat uptake. Based on a previous (unpublished) study from our group with a test / re-test design using18F-FTHA PET together with a mixed meal, we can estimate a sample size based on the repeatability coefficient (RCP) of 45% in visceral adipose tissue. With a significance level of 0.05 and power of 80% and, the investigators will need 10 individuals to detect a 15% difference in meal fat uptake in adipose tissue. In the event of participant dropout, additional individuals will be recruited to ensure the intended sample size is maintained.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes duration > 3 years or c-peptide negative
* Written and informed consent

Exclusion Criteria:

* Medicine with an impact on blood glucose or blood pressure
* Affected screening blood sample as evaluated by the clinical responsible investigator.
* Alcohol or substance abuse
* BMI > 35 kg/m2 or < 18.5 kg/m2
* Participation in other clinical trials involving ionized radiation within the last 6 months
* Lactose intolerance
* Doesn't speak and understand Danish.
* Severe claustrophobia.
* Commitment to special diets

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Difference in meal fat storage in visceral adipose tissue | 18F-FTHA PET scan 300 minutes after consumption of the liquid mixed meal
  Difference in meal fat storage (18F-FTHA PET scan) in visceral adipose tissue following a liquid mixed meal and varying the timing or skipping of meal insulin boluses.

SECONDARY OUTCOMES:
Difference in postprandial triglycerides | -20 to 360 minutes after consumption of the mixed meal
  Postprandial triglycerides measured as area under the curve ( iAUC of plasma triglyceride concentration).
Meal fat storage in target organs and tissues | 300 min after consumption of the mixed meal
  Differences in meal fat storage in skeletal muscle, liver, brain, and subcutaneous fat adipose tissue (18F-FTHA PET scan) following a mixed meal, comparing different timings of insulin administration.
Postprandial hormonal response and metabolites | -20 to 360 minutes after consumption of the mixed meal
  Plasma concentrations of free fatty acids, insulin, glucagon, blood glucose, and potentially others following a liquid test meal, comparing different timings of insulin administration.

CONTACTS AND LOCATIONS:
Overall Officials: Esben Søndergaard, MD, PhD, Study Director — Steno Diabetes Center Aarhus, Aarhus University Hospital, 8200 Aarhus, Denmark
Locations (1):
- Department of Nuclear Medicine & PET-Centre, AUH Palle Juul-Jensens Blvd. 165, 8200 Aarhus N, Denmark and Medical Research Laboratories/Steno Diabetes Center Aarhus, AUH Palle Juul-Jensens Blvd. 11, 8200 Aarhus N, Denmark, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No